CLINICAL TRIAL: NCT05998239
Title: Testing Bootle Boot Camp - A New Movement Tracking App to Engage Kids in Home Exercise Programs
Brief Title: Home Exercise Program Using Bootle Boot Camp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 0607
Record Dates: First submitted 2023-07-25; First posted 2023-08-18 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Our study is a semi-randomized, non-blinded single case experimental design with alternating treatments. The comparison period will consist of Bootle Boot Camp exercise sessions offered with movement tracking feedback alternating with exercise sessions offered without this feedback (4 sessions per week x 4 week). Children will be randomized to 1 of 16 alternating treatment schedules. The version of the App providing the most therapeutic data pattern will be used for an additional two weeks.
  We will also use a mixed methods sequential explanatory approach, with quantitative data collected in weeks 1-6 and qualitative data in weeks 7-8.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bootle Boot Camp with movement tracking feedback (virtual Coach Botley present) (Experimental): Bootle Boot Camp exercise sessions offered with movement tracking feedback through the presence of virtual coach Botley.
  Interventions: Other: Bootle Boot Camp Home Exercise App - with Virtual Coach Botley
- Bootle Boot Camp without movement tracking feedback (virtual Coach Botley absent) (Experimental): Bootle Boot Camp exercise sessions offered without movement tracking feedback through the absence of virtual coach Botley.
  Interventions: Other: Bootle Boot Camp Home Exercise App - without Virtual Coach Botley

INTERVENTIONS:
Other: Bootle Boot Camp Home Exercise App - with Virtual Coach Botley — Bootle Boot Camp exercise sessions offered with movement tracking feedback will be provided for a maximum of two consecutive sessions before being alternated with the no feedback condition for a period of 4 weeks (4 sessions/week). Movement feedback will be guided by skeletal data captured by the 3D motion tracking camera and based on predefined movement acceptability criteria for each exercise. Feedback will take the form of visual markers, text/audio cues and rewards.
  Arms: Bootle Boot Camp with movement tracking feedback (virtual Coach Botley present)
Other: Bootle Boot Camp Home Exercise App - without Virtual Coach Botley — Bootle Boot Camp exercise sessions offered without movement tracking feedback will be provided for a maximum of two consecutive sessions before being alternated with the movement tracking feedback condition for a period of 4 weeks (4 sessions/week).
  Arms: Bootle Boot Camp without movement tracking feedback (virtual Coach Botley absent)

SUMMARY:
This study aims to learn about the engagement and lower limb motor outcomes of children with cerebral palsy, ages 6-12 years, GMFCS Levels I-II, engaging in home-based movement practice using a novel therapy exercise Application, Bootle Boot Camp, offered with and without movement-tracking feedback.

DETAILED DESCRIPTION:
Adherence to home exercise programs is low. Interactive computer play (ICP) - any kind of computer game or virtual reality technology that allows users to interact with simulated objects in a virtual environment - offers a fun and motivational way to increase movement practice.

Bootle Boot Camp is a novel ICP technology developed by the Possibility Engineering and Research Lab at Holland Bloorview Kids Rehabilitation Hospital that uses a 3D motion tracking camera to provide real time feedback on skeletal movements during game play. It allows physiotherapists to prescribe personalized lower limb home exercise programs to clients.

The investigator's specific objectives are:

1. To compare participants' level of affective, behavioural, and cognitive engagement with Bootle Boot Camp with and without movement tracking feedback
2. To determine the quality of exercise performance when participants use Bootle Boot Camp with and without movement tracking feedback
3. To estimate the treatment response associated with use of Bootle Boot Camp
4. To explore physiotherapists, children, and their caregivers' experiences with the App.

Children with cerebral palsy (ages 6-12 years, GMFCS Level I or II) will be prescribed a home exercise program by their treating physiotherapist that they will complete independently using the App on their television at home. Bootle Boot Camp exercise sessions offered with movement-tracking feedback will be alternated with sessions offered without feedback for 4 weeks (4 sessions per week). Following this comparison period, the version of the App providing the most therapeutic data pattern based on system data and children's input will be used for an additional 2 weeks. Post 6 weeks of Bootle Boot Camp game play, children and caregivers will be asked to take part in semi-structured interviews to learn more about families' experiences with the home program

ELIGIBILITY:
Physiotherapist Inclusion Criteria:

* Registered and in good standing with the College of Physiotherapists of Ontario
* Minimum 1-year pediatric clinical experience
* Caseload consists of clients with cerebral palsy (ages 6-12 years; GMFCS Level I-II)
* Works in public sector (Holland Bloorview) or private sector (clinics) within Ontario
* Has technology (e.g., laptop) and internet services needed to use Bootle Boot Camp, complete online surveys and video calls
* Has managerial and institutional approval

Physiotherapist Exclusion Criteria:

* Visual/auditory deficits that would limit the physiotherapist's ability to interact with the App

Child Inclusion Criteria:

* Diagnosis of cerebral palsy (GMFCS Levels I-II)
* Ages 6-12 years
* Minimum 1 lower limb goal
* Able to complete 4 weekly exercise sessions using Bootle Boot Camp for 6 weeks
* Not currently receiving physiotherapy services more than once every two months (on an off block from physiotherapy)
* Normal or corrected to normal vision and hearing
* Child and parent can speak and understand English
* Has technology (e.g., laptop) and internet services needed to use Bootle Boot Camp, complete online surveys, and video calls
* Child's physiotherapist and parent able and willing to also participate in the study

Child Exclusion Criteria:

* Botox injection in the last 6 weeks or orthopedic surgery in the last 6 months
* Has serial casting, Botox injection, orthopedic surgery or other significant medical intervention during the 6-week training period with the App
* Photosensitivity or unstable epilepsy triggered by video games, screen activities or TV light
* Visual or auditory deficits that would limit gameplay
* Respiratory, cardiovascular, or other significant medical condition that would limit safe gameplay
* Engaging in a progressive lower limb muscle strengthening or balance home exercise program as prescribed by a health care provider
* An extensive medical or therapeutic schedule (services scheduled on more than 3 days/week)
* Scheduled event (e.g., family or school trip) that would limit ability to perform 4 sessions/week for 6 weeks during training period with the App

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Adherence (as a measure of behavioural engagement) | Week 1 - 6
  The number of exercise repetitions that are attempted each session will be tracked and recorded by the 3D camera computer system and will be expressed as a proportion of the total number of prescribed repetitions

SECONDARY OUTCOMES:
Smileyometer Scale | Week 1 - 6; Session 1 - 24
  Children will rate their level of fun and how helpful they feel the game is for their body after each exercise session using customized Smileyometer rating scales. The Smileyometer scale is a 5-point smiley face rating scale with anchors of 1 relating to "Awful" and 5 to "Brilliant" that is used to measure product liking. Higher scores reflect greater experienced fun.
Exercise fidelity | Week 1 - 6; Session 1 - 24
  The total acceptable repetition count (based on predefined movement quality criteria) for each exercise will be tracked and recorded by the 3D camera computer system and will be expressed as a proportion of the total number of prescribed repetitions.
Bootle Boot Camp Acceptability Survey | 4th week mark at session 16
  Children will rate perceived therapeutic effectiveness of each version of the App after the 4-week comparison period using the study-specific Bootle Boot Camp Acceptability Survey. The survey consists of questions with open-ended responses, rating agreement with statements (e.g., I had fun playing Bootle Boot Camp) on a 5-point rating scale with 1 representing 'disagree' to 5 representing 'agree,' and selecting which version of the App they feel best answers each question (e.g., which version of the game was most helpful for your body?)
Five Time Sit to Stand Test | Week 1 at session 1 & Week 6 at session 21
  The test measures the time needed to complete five consecutive sit to stand cycles as fast as possible as a measure of lower limb functional strength. Children will complete this test at the start and end of their six weeks of game play with Bootle Boot Camp
Modified Timed Up and Go | Week 1 at session 2 & Week 6 at session 22
  The test measures the time in seconds to rise from a chair, walk 3m and return to sitting as a measure of functional mobility. Children will complete this test at the start and end of their six weeks of game play with Bootle Boot Camp.
One Leg Stance Test | Week 1 at session 3 & Week 6 at session 23
  The test measures the time in seconds that a child can balance on one leg as a measure of standing stability. Children will complete this test at the start and end of their six weeks of game play with Bootle Boot Camp
Pediatric Reach Test | Week 1 at session 3 & Week 6 at session 23
  The test measures the distance that a child can reach forward and sideways in standing and sitting as a measure of balance. Children will complete this test at the start and end of their six weeks of game play with Bootle Boot Camp
30 Second Sit to Stand Test | Week 1 at session 4 & Week 6 at session 24
  The test measures the number of sit to stand cycles that a child can complete in 30 seconds as a measure of functional lower limb strength. Children will complete this test at the start and end of their six weeks of game play with Bootle Boot Camp
Mobile App Rating Scale | Week 4 at session 16
  Parents will complete the Mobile App Rating Scale (MARS) for each version of the game to assess each version's value and usability. The MARS assesses App quality through 5 subscales: engagement, functionality, aesthetics, information quality and subjective quality, with questions asked using 1-5 rating scales. An App quality mean score and App subjective quality score is reported. Higher scores denote more positive feelings towards the App.
Canadian Occupational Performance Measure | Week 0 and Week 7
  The Canadian Occupational Performance Measure (COPM) will be used to assess client's performance and satisfaction on self-identified goals pre and post six weeks of Bootle Boot Camp game play. Children rate performance and satisfaction on each activity using 10-point rating scales (minimum score 1 and maximum score 10) with higher scores reflecting higher performance and satisfaction. A change of at least 2 points has been considered clinically meaningful.
System Usability Scale and Bootle Boot Camp Usability Survey | Week 0
  Physiotherapists will rate the usability of Bootle Boot Camp using the System Usability Scale (SUS) after they have used the App to prescribe a home exercise program to their client. The SUS is composed of 10 questions with SUS scores ranging from 0 to 100, with higher scores reflecting greater usability.
Pick-A-Mood | Week 1 - 6; Session 1 - 24
  Before each exercise session, children will be asked how they are feeling using Pick-A-Mood, a cartoon-based self-report scale with eight characters representing eight different mood states.
Semi structured interviews | Week 7 and Week 8
  Children and parents will be interviewed post 6-weeks of Bootle Boot Camp game play to understand families' experiences with using the App for home exercise program completion
Wong-Bakers Faces Pain Scale | Week 1 - 6; Session 1 - 24
  Before each exercise session, children will be asked to rate their level of pain using the Wong Bakers Faces Pain scale, ranging from no pain (score of 0) to the most pain possible (score of 5). Higher scores denote more pain.
Study-specific Energy Level Question | Week 1 - 6; Session 1 - 24
  Before each exercise session, children will be asked to rate their level of energy using a study-specific energy level scale ranging from no energy (score of 0) to lots of energy (score of 10). Higher scores denote more energy.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, Principal Investigator — Bloorview Research Institute
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrevska M, Wright FV, Khan A, Munce S, Fehlings D, Biddiss E. Evaluating the impact of movement tracking feedback on engagement with home exercise programmes of children with cerebral palsy using a new therapy app: a protocol for a mixed-methods single-case experimental design with alternating treatments. BMJ Open. 2024 Mar 18;14(3):e082761. doi: 10.1136/bmjopen-2023-082761. PMID 38503423